CLINICAL TRIAL: NCT02094261
Title: Phase II, Open Label, Single-arm Study to Assess Safety and Efficacy of AZD9291 in Patients With Locally Advanced/Metastatic NSCLC Whose Disease Has Progressed With Previous EGFR TKI and Whose Tumours Are EGFR and T790M Mutation Positive
Brief Title: Phase II AZD9291 Open Label Study in NSCLC After Previous EGFR TKI Therapy in EGFR and T790M Mutation Positive Tumours
Acronym: AURA2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D5160C00002; 2014-000531-17 (EudraCT Number)
Record Dates: First submitted 2014-03-17; First posted 2014-03-21 (Estimated); Results first posted 2016-06-07 (Estimated); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Phase II, open label study; safety and efficacy of AZD9291; diagnosis of Epidermal Growth Factor Receptor mutation positive and T790M mutation positive NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AZD9291 (Experimental): Once daily tablet 80 mg
  Interventions: Drug: AZD9291

INTERVENTIONS:
Drug: AZD9291 — Once daily tablet 80 mg

SUMMARY:
A Phase II, Open Label, Single-arm Study to Assess the Safety and Efficacy of AZD9291 in Patients with Locally Advanced/Metastatic Non Small Cell Lung Cancer whose Disease has Progressed with Previous Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitor Therapy and whose Tumours are Epidermal Growth Factor Receptor Mutation and T790M Mutation Positive

DETAILED DESCRIPTION:
This is a phase II, open label, single arm study assessing the safety and efficacy of AZD9291 (80 mg, orally, once daily) in patients with a confirmed diagnosis of Epidermal Growth Factor Receptor mutation positive and T790M mutation positive NSCLC,who have progressed following prior therapy with an approved Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitor (EGFR-TKI) agent. Patients must agree to provide a biopsy for central confirmation of T790M mutation status following confirmed disease progression on the most recent treatment regimen. The primary objective of the study is to assess the efficacy of AZD9291 by assessment of Objective Response Rate according to RECIST 1.1 by an Independent Central Review.

ELIGIBILITY:
Inclusion:

* Aged at least 18 years. Japan patients aged at least 20 years.
* Locally advanced/metastatic NSCLC not amenable to curative surgery or radiotherapy
* Radiological documentation of disease progression:

following 1st line EGFR TKI treatment but who have not received further treatment OR following prior therapy with an EGFR TKI and a platinum-based doublet chemotherapy. Patients who received prior EGFR TKI and platinum-based doublet chemotherapy may have also received additional lines of treatment. All patients must have documented radiological progression on the last treatment administered prior to enrolling in the study.

* Disease progression following 1st line EGFR TKI treatment or following prior EGFR TKI and platinum-containing doublet chemotherapy.
* Confirmation that the tumour harbours an EGFR mutation known to be associated with EGFR TKI sensitivity (including G719X, exon 19 deletion, L858R, L861Q). Patients must have central confirmation of tumour T790M mutation positive status from a biopsy sample taken after confirmation of disease progression on the most recent treatment regimen.
* World Health Organisation (WHO) performance status 0-1 with no deterioration over the previous 2 weeks and a minimum life expectancy of 12 weeks.
* At least one lesion, not previously irradiated and not chosen for biopsy during the study screening period, that can be accurately measured at baseline as ≥ 10mm in the longest diameter (except lymph nodes which must have short axis ≥ 15mm) with computerised tomography (CT) or magnetic resonance imaging (MRI) which is suitable for accurate repeated measurements.
* Females of child-bearing potential using contraception; negative pregnancy test.

Exclusion:

* Treatment with an EGFR-TKI within 8 days of study entry; any cytotoxic chemotherapy, investigational agents or other anticancer drugs within 14 days of study entry; previous treatment with AZD9291 (or 3rd generation TKIs); major surgery within 4 weeks; radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation within 4 weeks; current treatment with potent inhibitors of CYP2C8 and potent inhibitors/inducers of CYP3A4.
* Unresolved toxicities from prior therapy.
* Unstable spinal cord compression/brain metastases.
* Severe/uncontrolled systemic diseases, including uncontrolled hypertension, bleeding diatheses or infection.
* Refractory nausea/vomiting, chronic gastrointestinal diseases or bowel resection.
* Cardiac disease.
* Past history of ILD, drug-induced ILD, radiation pneumonitis which required steroid treatment, or any evidence of clinically active interstitial lung disease.
* Inadequate bone marrow reserve or organ function.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2014-05-20 (Actual); Primary Completion 2015-05-01 (Actual); Study Completion 2023-11-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Glenwood Goss, MD, Principal Investigator — 501 Smyth Road, Ottawa, Canada; Tetsuya Mitsudomi, MD, Principal Investigator — Kinki University Hospital, Faculty of Medicine, Osaka, Japan
Locations (41):
- United States (9):
  - Research Site, La Jolla, California
  - Research Site, Orange, California
  - Research Site, New Haven, Connecticut
  - Research Site, Norwalk, Connecticut
  - Research Site, Indianapolis, Indiana
  - Research Site, Boston, Massachusetts
  - Research Site, Lebanon, New Hampshire
  - Research Site, New York, New York
  - Research Site, Durham, North Carolina
- Canada (3):
  - Research Site, Edmonton, Alberta
  - Research Site, Ottawa, Ontario
  - Research Site, Toronto, Ontario
- Hong Kong (2):
  - Research Site, Hong Kong
  - Research Site, Shatin
- Italy (4):
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Perugia
  - Research Site, Verona
- Japan (12):
  - Research Site, Akashi-shi
  - Research Site, Chūōku
  - Research Site, Kitaadachi-gun
  - Research Site, Kitakyushu-shi
  - Research Site, Kōtoku
  - Research Site, Nagoya
  - Research Site, Niigata
  - Research Site, Osaka
  - Research Site, Sakaishi
  - Research Site, Sayama
  - Research Site, Wakayama
  - Research Site, Yokohama
- South Korea (3):
  - Research Site, Goyang-si
  - Research Site, Seongnam-si
  - Research Site, Seoul
- Spain (6):
  - Research Site, A Coruña
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Majadahonda
  - Research Site, Málaga
  - Research Site, Valencia
- Taiwan (2):
  - Research Site, Taichung
  - Research Site, Taipei

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Murat-Onana ML, Ramalingam SS, Janne PA, Gray JE, Ahn MJ, John T, Yatabe Y, Huang X, Rukazenkov Y, Javey M, Brown H, Li-Sucholeiki X. EGFR mutation testing across the osimertinib clinical program. Lung Cancer. 2025 Jun;204:108549. doi: 10.1016/j.lungcan.2025.108549. Epub 2025 Apr 18. PMID 40311309
- [Derived] Ahn MJ, Han JY, Kim DW, Cho BC, Kang JH, Kim SW, Yang JC, Mitsudomi T, Lee JS. Osimertinib in Patients with T790M-Positive Advanced Non-small Cell Lung Cancer: Korean Subgroup Analysis from Phase II Studies. Cancer Res Treat. 2020 Jan;52(1):284-291. doi: 10.4143/crt.2019.200. Epub 2019 Jul 23. PMID 31345012
- [Derived] Ahn MJ, Tsai CM, Shepherd FA, Bazhenova L, Sequist LV, Hida T, Yang JCH, Ramalingam SS, Mitsudomi T, Janne PA, Mann H, Cantarini M, Goss G. Osimertinib in patients with T790M mutation-positive, advanced non-small cell lung cancer: Long-term follow-up from a pooled analysis of 2 phase 2 studies. Cancer. 2019 Mar 15;125(6):892-901. doi: 10.1002/cncr.31891. Epub 2018 Dec 4. PMID 30512189
- [Derived] Goss G, Tsai CM, Shepherd FA, Ahn MJ, Bazhenova L, Crino L, de Marinis F, Felip E, Morabito A, Hodge R, Cantarini M, Johnson M, Mitsudomi T, Janne PA, Yang JC. CNS response to osimertinib in patients with T790M-positive advanced NSCLC: pooled data from two phase II trials. Ann Oncol. 2018 Mar 1;29(3):687-693. doi: 10.1093/annonc/mdx820. PMID 29293889
- [Derived] Goss G, Tsai CM, Shepherd FA, Bazhenova L, Lee JS, Chang GC, Crino L, Satouchi M, Chu Q, Hida T, Han JY, Juan O, Dunphy F, Nishio M, Kang JH, Majem M, Mann H, Cantarini M, Ghiorghiu S, Mitsudomi T. Osimertinib for pretreated EGFR Thr790Met-positive advanced non-small-cell lung cancer (AURA2): a multicentre, open-label, single-arm, phase 2 study. Lancet Oncol. 2016 Dec;17(12):1643-1652. doi: 10.1016/S1470-2045(16)30508-3. Epub 2016 Oct 14. PMID 27751847
- See also: D5160C00002_12_1_01csp_andamendments_Redacted1 — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1881&filename=D5160C00002_12_1_01csp_andamendments-redaction_proposal_Redacted1.pdf
- See also: CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5160C00002&attachmentIdentifier=97782bed-6ea3-43cb-a776-b78794b0b1a4&fileName=d5160c00002-study-synopsis_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient enrolled: 28 April 2014, Data cut off: 1 May 2015. The study was open for enrolment at 44 study centres in Canada (3), Hong Kong (2), Italy (5), Japan (14), South Korea (3), Spain (6), Taiwan (2), and the USA (9). Recruitment has closed and primary analyses have been performed but study is still on-going.
Pre-assignment Details: 472 patients were enrolled (signed informed consent). Patients were assigned to treatment if they met all the inclusion and none of the exclusion criteria. 262 patients were enrolled but failed inclusion/exclusion criteria and so were not eligible to be assigned treatment. The remaining 210 patients received treatment.
Groups:
- AZD9291 80mg: Daily single dose of AZD9291 80mg
Period: Overall Study
Arm/Group | AZD9291 80mg
Started | 210
Completed | 0
Not Completed | 210
Not completed — Death | 24
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 4
Not completed — Ongoing Study at Data Cut-off | 181

BASELINE CHARACTERISTICS:
Arm/Group | AZD9291 80mg
Number analyzed (Participants) | 210
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.9 (10.91) [35 to 88]
Age, Customized [Number; unit: Participants]
  <50 Years | 20
  >=50-<65 Years | 88
  >=65-<75 Years | 69
  >=75 Years | 33
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 146
  Male | 64
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 132
  Black Or African American | 3
  Native Hawaiian Or Other Pacific Islander | 1
  Other | 2
  White | 72

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: Per Response Evaluation Criteria in Solid Tumours (RECIST v1.1) assessed by MRI or CT: Complete Response (CR): Disappearance of all target and non-target lesions and no new lesions; Partial Response (PR): >= 30% decrease in the sum of diameters of Target Lesions (compared to baseline) and no new lesions. ORR is the percentage of patients with at least 1 visit response of CR or PR (according to independent review) that was confirmed at least 4 weeks later, prior to progression or further anti-cancer therapy.
Time Frame: RECIST tumour assessments every 6 weeks from first dose until objective disease progression, up to approximately 11 months (at the time of analysis)
Population: All patients who received at least 1 dose of study treatment and had measurable disease at baseline according to the independent review of baseline imaging data.
Measure: Number (95% Confidence Interval); unit: % of participants
Arm/Group | AZD9291 80mg
Number analyzed (Participants) | 199
% of participants | 70.9 [64.0 to 77.1]

2. Secondary Outcome: Duration of Response (DoR)
Description: Per Response Evaluation Criteria in Solid Tumours (RECIST v1.1) assessed by MRI or CT: Complete Response (CR): Disappearance of all target and non-target lesions and no new lesions; Partial Response (PR): >= 30% decrease in the sum of diameters of Target Lesions (compared to baseline) and no new lesions. DoR was defined as the time from the date of first documented response (CR or PR that was subsequently confirmed) until the date of documented progression (PD) or death in the absence of disease progression (by investigator assessment).
Time Frame: as for outcome 1
Population: All patients who received at least 1 dose of study treatment, had measurable disease at baseline according to the independent review of baseline imaging data and had confirmed response.
Measure: Median (Full Range); unit: months
Arm/Group | AZD9291 80mg
Number analyzed (Participants) | 141
months | 7.8 [1.3 to 8.4]

3. Secondary Outcome: Disease Control Rate (DCR)
Description: Per Response Evaluation Criteria in Solid Tumours (RECIST v1.1) assessed by MRI or CT: Complete Response (CR): Disappearance of all target and non-target lesions and no new lesions; Partial Response (PR): >= 30% decrease in the sum of diameters of Target Lesions (compared to baseline) and no new lesions; Stable disease (SD): Neither sufficient shrinkage to qualify as a response nor sufficient growth to qualify as progression; Progressive Disease (PD): >= 20% increase in the sum of diameters of TLs and an absolute increase in sum of diameters of >=5mm (compared to the previous minimum sum) or progression of NTLs or a new lesion. DCR is the percentage of patients with best response of CR, PR or SD (according to independent review), prior to progression (PD) or further anti-cancer therapy.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: % of participants
Arm/Group | AZD9291 80mg
Number analyzed (Participants) | 199
% of participants | 91.5 [86.7 to 94.9]

4. Secondary Outcome: Progression-Free Survival (PFS)
Description: Per Response Evaluation Criteria in Solid Tumours (RECIST v1.1) assessed by MRI or CT: Progressive Disease (PD): >= 20% increase in the sum of diameters of TLs and an absolute increase in sum of diameters of >=5mm (compared to the previous minimum sum) or progression of NTLs or a new lesion. PFS is the time from date of first dose until the date of PD (by independent review) or death (by any cause in the absence of progression) regardless of whether the patient withdrew from AZD9291 therapy or received another anti-cancer therapy prior to progression. Patients who had not progressed or died at the time of analysis were censored at the time of the latest date of assessment from their last evaluable RECIST 1.1 assessment.
Time Frame: as for outcome 1
Population: All patients who received at least 1 dose of study treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | AZD9291 80mg
Number analyzed (Participants) | 210
months | 8.6 [8.28 to 9.72]

ADVERSE EVENTS:
Time Frame: AEs from start of study drug until 28 days post treatment discontinuation, up to approximately 11 months (at time of analysis).
Description: Systematic assessment due to regular investigator assessment at study visits.
Arm/Group | AZD9291 80mg
Serious Adverse Events (participants affected / at risk) | 42/210
Other Adverse Events (participants affected / at risk) | 193/210
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD9291 80mg (N=210)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 2 (2)
Hearing impaired (Ear and labyrinth disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Pharyngeal abscess (Infections and infestations) | 1 (2)
Pneumonia (Infections and infestations) | 4 (5)
Sepsis (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Radiation necrosis (Injury, poisoning and procedural complications) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1)
Cerebral infarction (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 8 (9)
Deep vein thrombosis (Vascular disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD9291 80mg (N=210)
Anaemia (Blood and lymphatic system disorders) | 19 (19)
Thrombocytopenia (Blood and lymphatic system disorders) | 11 (15)
Dry eye (Eye disorders) | 11 (11)
Abdominal pain upper (Gastrointestinal disorders) | 11 (14)
Constipation (Gastrointestinal disorders) | 32 (38)
Diarrhoea (Gastrointestinal disorders) | 81 (115)
Nausea (Gastrointestinal disorders) | 34 (35)
Stomatitis (Gastrointestinal disorders) | 22 (31)
Vomiting (Gastrointestinal disorders) | 16 (18)
Asthenia (General disorders) | 11 (12)
Fatigue (General disorders) | 31 (33)
Oedema peripheral (General disorders) | 17 (18)
Nasopharyngitis (Infections and infestations) | 21 (23)
Paronychia (Infections and infestations) | 32 (32)
Upper respiratory tract infection (Infections and infestations) | 11 (11)
Urinary tract infection (Infections and infestations) | 13 (16)
Alanine aminotransferase increased (Investigations) | 15 (17)
Aspartate aminotransferase increased (Investigations) | 12 (12)
Electrocardiogram QT prolonged (Investigations) | 11 (13)
Neutrophil count decreased (Investigations) | 14 (17)
Platelet count decreased (Investigations) | 20 (23)
White blood cell count decreased (Investigations) | 16 (22)
Decreased appetite (Metabolism and nutrition disorders) | 29 (32)
Arthralgia (Musculoskeletal and connective tissue disorders) | 18 (19)
Back pain (Musculoskeletal and connective tissue disorders) | 25 (26)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 11 (11)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 14 (15)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 14 (14)
Dizziness (Nervous system disorders) | 11 (11)
Headache (Nervous system disorders) | 20 (25)
Insomnia (Psychiatric disorders) | 11 (11)
Cough (Respiratory, thoracic and mediastinal disorders) | 25 (31)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 14 (16)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 16 (16)
Dry skin (Skin and subcutaneous tissue disorders) | 52 (58)
Pruritus (Skin and subcutaneous tissue disorders) | 32 (33)
Rash (Skin and subcutaneous tissue disorders) | 49 (58)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 14 (17)
Skin fissures (Skin and subcutaneous tissue disorders) | 12 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 180 days from the time submitted to the sponsor for review, should the submission for publication be delayed in order to file patent application. The sponsor cannot require changes to the communication and cannot extend the embargo.